CLINICAL TRIAL: NCT01158222
Title: A Phase II Study of Intermittent Sunitinib in Previously Untreated Patients With Metastatic Renal Cell Carcinoma
Brief Title: Sunitinib Malate in Treating Patients With Previously Untreated Metastatic Kidney Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Case Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CASE8809; NCI-2010-01391 (Other: NCI/CTRP)
Record Dates: First submitted 2010-07-06; First posted 2010-07-08 (Estimated); Results first posted 2018-08-16 (Actual); Last update posted 2018-09-14 (Actual); Status verified 2018-08

CONDITIONS: Clear Cell Renal Cell Carcinoma; Stage IV Renal Cell Cancer
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — Sunitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Arm I (Experimental): Patients receive oral sunitinib malate once daily on days 1-28. Treatment repeats every 42 days for at least 4 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: sunitinib malate

INTERVENTIONS:
Drug: sunitinib malate — Given orally
  Other Names: SU011248; SU11248; sunitinib; Sutent

SUMMARY:
RATIONALE: Sunitinib malate may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth or by blocking blood flow to the tumor.

PURPOSE: This phase II trial is studying how well sunitinib malate it works in treating patients with previously untreated metastatic kidney cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the feasibility of intermittent sunitinib therapy in patients with metastatic renal cell carcinoma (RCC).

SECONDARY OBJECTIVES:

I. To determine the clinical outcome (response rate and overall progression-free survival) in metastatic renal cell carcinoma patients treated with intermittent sunitinib therapy.

II. To evaluate the toxicity of intermittent sunitinib therapy in patients with metastatic renal cell carcinoma.

III. To assess the feasibility of detecting circulating tumor cells (CTCs) in RCC patients and investigate the association between the VEGF -634 genotype and the occurrence of hypertension in sunitinib-treated RCC patients.

OUTLINE:

Patients receive oral sunitinib malate once daily on days 1-28. Sunitinib dosing schedule may be changed to 14 days on followed by 7 days off, and repeated for a 6-week cycle, at the discretion of the treating physician for toxicity purposes. Cycles will be defined as 6 week intervals regardless of dosing interruptions. All patients will be treated for 4 cycles in the absence of unacceptable toxicity or RECIST-defined progressive disease.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically-proven advanced RCC with a component of clear cell histology
* Measurable disease per RECIST criteria
* ECOG performance status 0-1
* Prior nephrectomy is NOT required
* Serum aspartate transaminase (AST; serum glutamic oxaloacetic transaminase [SGOT]) and serum alanine transaminase (ALT; serum glutamic pyruvic transaminase [SGPT]) ≤ 2.5 x laboratory upper limit of normal (ULN)
* Total serum bilirubin ≤ 2.0 x ULN
* Absolute neutrophil count (ANC) ≥ 1500/uL
* Platelets ≥ 100,000/uL
* Hemoglobin ≥ 8.0 g/dL (transfusion permitted)
* Serum calcium ≤ 12.0 mg/dL
* Serum creatinine ≤ 2.5 mg/dL
* Patients with history of brain metastases can be enrolled at a minimum of 2 weeks following the completion of surgery, gamma knife or whole brain radiotherapy; repeat brain MRI not required for eligibility
* Signed and dated informed consent document indicating that the patient (or legally acceptable representative) has been informed of all pertinent aspects of the trial prior to enrollment

Exclusion Criteria:

* Prior systemic treatment for advanced RCC. Prior adjuvant therapy (any drug) is allowed if end of adjuvant therapy was more than 1 year prior to start of sunitinib on this protocol.
* Any of the following within the 6 months prior to study drug administration: myocardial infarction, severe/unstable angina, severe peripheral vascular disease (claudication) or procedure on peripheral vasculature, coronary/peripheral artery bypass graft, New York Heart Association grade II or greater congestive heart failure, cerebrovascular accident or transient ischemic attack, clinically significant bleeding or pulmonary embolism
* Hypertension that cannot be controlled by medications to < 160/90 mmHg
* Known human immunodeficiency virus (HIV) or acquired immunodeficiency syndrome (AIDS)-related illness
* Pregnancy or breastfeeding
* Other severe acute or chronic medical or psychiatric conditions or laboratory abnormality that may increase the risk associated with study participation or study drug administration, or may interfere with the interpretation of study results, and in the judgment of the investigator would make the patient inappropriate for entry into this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2010-08-18 (Actual); Primary Completion 2013-06-20 (Actual); Study Completion 2017-02-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brian Rini, Principal Investigator — Cleveland Clinic Taussig Cancer Institute, Case Comprehensive Cancer Center
Locations (1):
- Cleveland Clinic Taussig Cancer Institute, Case Comprehensive Cancer Center, Cleveland, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 5 additional patients were consented but not enrolled in the study. No information was collected on them and they are not included in the patient flow. Demographics information was not collected on these patients.
Groups:
- Arm I: Patients receive oral sunitinib malate once daily on days 1-28. Treatment repeats every 42 days for at least 4 courses in the absence of disease progression or unacceptable toxicity.
  sunitinib malate: Given orally
  laboratory biomarker analysis: Correlative studies
  reverse transcriptase-polymerase chain reaction: Correlative studies
  polymorphism analysis: Correlative studies
Period: Overall Study
Arm/Group | Arm I
Started | 37
Completed | 20
Not Completed | 17
Not completed — Not eligible for intermediate phase | 17

BASELINE CHARACTERISTICS:
Arm/Group | Arm I
Number analyzed (Participants) | 37
Age, Customized [Count of Participants; unit: Participants]
  40-49 | 3
  50-59 | 9
  60-69 | 18
  70-79 | 6
  80-89 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 26
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 35
  Unknown or Not Reported | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 34
  More than one race | 0
  Unknown or Not Reported | 2
Region of Enrollment [Number; unit: participants]
  United States | 37

OUTCOME MEASURES:

1. Primary Outcome: Feasibility as Assessed by Proportion of Patients Eligible for Intermittent Therapy Who Actually Receive it
Description: Treatment repeats every 42 days for at least 4 courses in the absence of disease progression or unacceptable toxicity.
Time Frame: after 6 months of treatment (4 cycles)
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I
Number analyzed (Participants) | 20
Participants | 20

2. Secondary Outcome: Change in Circulating Tumor Cells
Time Frame: Pre-treatment, day 1, and day 28 of every cycle
Population: Did not complete this analysis. Data not collected.
Arm/Group | Arm I
Number analyzed (Participants) | 0

3. Secondary Outcome: Relationship Between Hypertension and Germline VEGF Single Nucleotide Polymorphism (SNP) -634 Genotype
Time Frame: Day 28 of each cycle
Population: Did not complete this analysis. Data not collected.
Arm/Group | Arm I
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | Arm I
All-Cause Mortality (participants affected / at risk) | 2/37
Serious Adverse Events (participants affected / at risk) | 13/37
Other Adverse Events (participants affected / at risk) | 37/37
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (N=37)
Atrial Fibrillation (Cardiac disorders) | 1 (1)
Abdominal Pain (Gastrointestinal disorders) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Gastrointestinal disorder - other (Gastrointestinal disorders) | 1 (1) — GI bleeding
Chills (General disorders) | 1 (1)
Edema Trunk (General disorders) | 1 (1) — lower extremity edema
Fever (General disorders) | 1 (1)
Abdominal infection (Infections and infestations) | 1 (1)
Infection and infestation - other (Infections and infestations) | 1 (1) — Infection
Lung infection (Infections and infestations) | 1 (1)
Upper respiratory infection (Infections and infestations) | 2 (2)
Urinary tract infection (Infections and infestations) | 1 (1)
Weight Gain (Investigations) | 1 (1)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (1)
Intracranial Hemorrhage (Nervous system disorders) | 1 (1)
Syncope (Nervous system disorders) | 1 (2)
Hematuria (Renal and urinary disorders) | 1 (1)
Proteinuria (Renal and urinary disorders) | 1 (1)
Renal and urinary disorders - other (Renal and urinary disorders) | 1 (1) — death from metastatic renal cancer
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Respiratory, thoracic and mediastinal disorders - other (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Pneumonia
Palmar-Plantar Erythrodysesthesia Syndrome (Skin and subcutaneous tissue disorders) | 1 (1) — Hand-Foot Syndrome
Thromboembolic Event (Vascular disorders) | 1 (1) — pulmonary embolism
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (N=37)
Anemia (Blood and lymphatic system disorders) | 26 (67)
Blood and lymphatic system disorders - other (Blood and lymphatic system disorders) | 2 (2) — erythrocytosis
Hyperthyroidism (Endocrine disorders) | 3 (3)
Hypothyroidism (Endocrine disorders) | 18 (24)
Abdominal distension (Gastrointestinal disorders) | 2 (2)
Abdominal Pain (Gastrointestinal disorders) | 9 (12)
Cheilitis (Gastrointestinal disorders) | 4 (7)
Constipation (Gastrointestinal disorders) | 18 (32)
Dental Caries (Gastrointestinal disorders) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 23 (88)
Dry Mouth (Gastrointestinal disorders) | 4 (5)
Dyspepsia (Gastrointestinal disorders) | 19 (35)
Flatulence (Gastrointestinal disorders) | 3 (4)
Gastroesophageal Reflux Disease (Gastrointestinal disorders) | 5 (6)
Gastrointestinal Disorders - Other (Gastrointestinal disorders) | 4 (9) — Early Satiety
Hemorrhoidal hemorrhage (Gastrointestinal disorders) | 6 (6)
Hemorrhoids (Gastrointestinal disorders) | 7 (7)
Lip Pain (Gastrointestinal disorders) | 2 (2)
Mucositis Oral (Gastrointestinal disorders) | 31 (107)
Nausea (Gastrointestinal disorders) | 25 (75)
Oral Hemorrhage (Gastrointestinal disorders) | 3 (3)
Oral Pain (Gastrointestinal disorders) | 3 (5)
Vomiting (Gastrointestinal disorders) | 13 (25)
Chills (General disorders) | 3 (5)
Edema limbs (General disorders) | 11 (15)
Fatigue (General disorders) | 35 (127)
Fever (General disorders) | 4 (8)
General Disorders - Other (General disorders) | 4 (4) — cold intolerance
Localized Edema (General disorders) | 2 (3)
Pain (General disorders) | 15 (35)
Lung Infection (Infections and infestations) | 2 (2)
Mucosal Infection (Infections and infestations) | 2 (3)
Nail Infection (Infections and infestations) | 2 (2)
Pharyngitis (Infections and infestations) | 3 (3)
Rhinitis Infective (Infections and infestations) | 2 (2)
Skin Infection (Infections and infestations) | 2 (9)
Tooth Infection (Infections and infestations) | 2 (4)
Upper Respiratory Infection (Infections and infestations) | 5 (6)
Urinary Tract Infection (Infections and infestations) | 4 (5)
Bruising (Injury, poisoning and procedural complications) | 3 (6)
Alanine Aminotransferase Increased (Investigations) | 10 (18)
Alkaline Phosphatase Increased (Investigations) | 3 (5)
Aspartate Aminotranferase Increased (Investigations) | 13 (34)
Blood Bilirubin Increased (Investigations) | 4 (7)
Creatinine Increased (Investigations) | 17 (39)
Lymphocyte Count Decreased (Investigations) | 4 (6)
Neutrophil Count Decreased (Investigations) | 18 (57)
Platelet Count Decreased (Investigations) | 31 (115)
Weight Gain (Investigations) | 3 (6)
Weight Loss (Investigations) | 14 (16)
White Blood Cell Decreased (Investigations) | 25 (73)
Anorexia (Metabolism and nutrition disorders) | 19 (53)
Dehydration (Metabolism and nutrition disorders) | 5 (5)
Hypercalcemia (Metabolism and nutrition disorders) | 2 (3)
Hyperclycemia (Metabolism and nutrition disorders) | 8 (18)
Hyperkalemia (Metabolism and nutrition disorders) | 6 (11)
Hyperuricemia (Metabolism and nutrition disorders) | 3 (5)
Hypoalbuminemia (Metabolism and nutrition disorders) | 5 (12)
Hypocalcemia (Metabolism and nutrition disorders) | 2 (4)
Hypokalemia (Metabolism and nutrition disorders) | 2 (4)
Hypomagnesemia (Metabolism and nutrition disorders) | 4 (4)
Hyponatremia (Metabolism and nutrition disorders) | 10 (32)
Hypophosphatemia (Metabolism and nutrition disorders) | 5 (5)
Arthralgia (Musculoskeletal and connective tissue disorders) | 9 (121)
Arthritis (Musculoskeletal and connective tissue disorders) | 2 (3)
Back Pain (Musculoskeletal and connective tissue disorders) | 5 (5)
Generalized Muscle Weakness (Musculoskeletal and connective tissue disorders) | 4 (11)
Muscle Weakness Lower Limb (Musculoskeletal and connective tissue disorders) | 2 (3)
Myalgia (Musculoskeletal and connective tissue disorders) | 9 (20)
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 11 (17)
Cognitive Disturbance (Nervous system disorders) | 4 (4)
Dizziness (Nervous system disorders) | 6 (6)
Dysgeusia (Nervous system disorders) | 26 (58)
Headache (Nervous system disorders) | 10 (21)
Syncope (Nervous system disorders) | 2 (2)
Anxiety (Psychiatric disorders) | 4 (4)
Depression (Psychiatric disorders) | 5 (6)
Insomnia (Psychiatric disorders) | 3 (3)
Hematuria (Renal and urinary disorders) | 2 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 7 (9)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 7 (12)
Sore Throat (Respiratory, thoracic and mediastinal disorders) | 2 (5)
Voice Alteration (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Alopecia (Skin and subcutaneous tissue disorders) | 4 (4)
Dry Skin (Skin and subcutaneous tissue disorders) | 14 (22)
Erythema Multiforme (Skin and subcutaneous tissue disorders) | 6 (11)
Erythroderma (Skin and subcutaneous tissue disorders) | 2 (2)
Pain of Skin (Skin and subcutaneous tissue disorders) | 4 (5)
Palmar-plantar Erythrodysesthesia Syndrome (Skin and subcutaneous tissue disorders) | 20 (78) — hand and foot syndrome
Pruritus (Skin and subcutaneous tissue disorders) | 8 (13)
Purpura (Skin and subcutaneous tissue disorders) | 8 (18)
Rash Acneiform (Skin and subcutaneous tissue disorders) | 10 (19)
Scalp Pain (Skin and subcutaneous tissue disorders) | 2 (2)
Skin and Subcutaneous Tissue Disorders - Other (Skin and subcutaneous tissue disorders) | 4 (12) — desquamation
Skin and Subcutaneous Tissue Disorders - Other (Skin and subcutaneous tissue disorders) | 6 (10) — skin color change
Hot Flashes (Vascular disorders) | 3 (3)
Hypertension (Vascular disorders) | 22 (45)
Bone Pain (Musculoskeletal and connective tissue disorders) | 3 (8)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes